CLINICAL TRIAL: NCT06629272
Title: Optimizing Care for Older Adults Through Thyroid Hormone Deprescribing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Maria Papaleontiou, Associate Professor of Internal Medicine and Research Associate Professor at the Institute of Gerontology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HUM00231965; 1R01AG079833-01A1 (NIH)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Hypothyroidism
Keywords: thyroid hormone overtreatment and misuse; older adults; deprescribing
MeSH Terms: conditions — Hypothyroidism | interventions — Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Because the intervention is educational in nature, blinding is not possible. But, to preserve a certain level of blinding and protect against bias, the study will be presented as a "medication optimization study" and consenting patient participants will be informed that their medication profiles will be transmitted to the research team within the following months and that they will receive a customized brochure at some point during the next year that may contain recommendations for change which they can discuss with their prescribing provider. For providers, blinding will be achieved by presenting the same study timeline. Providers will be aware that they will receive a customized letter with thyroid hormone optimization recommendations and that their patients will receive an intervention at some point during the following year, and remain blinded to group allocation throughout the course of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-THIO (Deprescribing Thyroid Hormone In Older Adults) (Experimental): D-THIO is an innovative adapted multilevel intervention.
  Providers in the intervention arm will receive: 1) an introductory letter, and 2) the D-THIO pharmaceutical opinion via EMR-compatible correspondence.
  After randomization of their treating providers, patients in the intervention arm will receive a study packet including: 1) introductory letter, and 2) the D-THIO patient brochure (educational EMPOWER brochure).
  Interventions: Behavioral: D-THIO (Deprescribing Thyroid Hormone In Older Adults)
- Enhanced usual care (Active Comparator): This arm will receive enhanced usual care.
  Providers in the control arm will receive: 1) an introductory letter signed by the PI and site-PIs, and 2) the ATA hypothyroidism pocket card via EMR.
  Patients in the control arm will receive a study packet including: 1) introductory letter, and 2) the ATA patient brochure.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: D-THIO (Deprescribing Thyroid Hormone In Older Adults) — D-THIO consists of evidence-based pharmaceutical opinion letters to providers advising deprescribing for their patients 65 years and older with thyroid hormone overtreatment/misuse and EMPOWER ("Eliminating Medications through Patient Ownership of End Results") brochures to their patients.
  Arms: D-THIO (Deprescribing Thyroid Hormone In Older Adults)
Behavioral: Enhanced usual care — American Thyroid Association [ATA] provider guidelines, ATA patient brochure
  Arms: Enhanced usual care

SUMMARY:
The proposed study focuses on testing a novel adapted evidence-based multilevel intervention, Deprescribing Thyroid Hormone In Older Adults (D-THIO), to support thyroid hormone deprescribing (dose de-escalation and/or discontinuation) in older adults with thyroid hormone overtreatment and/or misuse and reduce patient harm. Findings from this study will lay the groundwork for broad implementation of D-THIO and serve as a model for deprescribing inappropriate medications for other endocrine conditions and conditions with biochemical monitoring.

DETAILED DESCRIPTION:
The proposed study is the first multi-site trial to evaluate a novel evidence-based adapted multilevel intervention, D-THIO (Deprescribing Thyroid Hormone In Older Adults), consisting of evidence-based pharmaceutical opinion to providers, education brochures to patients and facilitated by clinical champions, to support thyroid hormone deprescribing in older adults. We will conduct a type 1 hybrid effectiveness-implementation trial of D-THIO vs. enhanced usual care (American Thyroid Association [ATA] provider abbreviated guidelines, ATA patient brochure) at 3 sites (University of Michigan, Henry Ford, University of California San Francisco) in 150 providers (primary care, endocrinologists, geriatricians, advance practice providers) and 750 of their patients 65 years and older who are overtreated with thyroid hormone. We will randomize 1:1 at the provider level within each site. The aims of the study are: 1) to assess the effectiveness of D-THIO on thyroid hormone deprescribing by providers and on reducing overtreatment and misuse with thyroid hormone via EMR, 2) to assess the effectiveness of D-THIO on provider and patient knowledge and attitudes regarding thyroid hormone deprescribing via surveys, and 3) to identify factors related to the implementation of D-THIO across diverse general care settings via post-trial interviews with key stakeholders.

ELIGIBILITY:
Patient Eligibility:

Inclusion Criteria:

1. age 65 years and older
2. on thyroid hormone therapy and have a serum Thyroid-stimulating hormone (TSH) <0.5 mIU/L or are on thyroid hormone therapy for an inappropriate indication
3. English speaking
4. without cognitive impairment

Exclusion Criteria:

1) Patients with a diagnosis of thyroid cancer, secondary hypothyroidism, history of total thyroidectomy or hospitalization in the past 3 months will be excluded.

Provider eligibility:

Inclusion: Primary care physicians, endocrinologists, geriatricians, and Advanced Practice Providers (APPs) who practice at University of Michigan, Henry Ford Health System or University of California San Fransico (UCSF) and who prescribe thyroid hormone for eligible patients identified above will be eligible for study participation.

Exclusion: Providers who don't prescribe thyroid hormone.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Thyroid hormone deprescribing by providers | 6 months post-enrollment
  Assessed by proportion of patients who had any thyroid hormone dose de-escalation and/or thyroid hormone discontinuation. Thyroid hormone deprescribing is defined as thyroid hormone dose de-escalation and/or discontinuation and will be assessed via Electronic Medical Record (EMR).

SECONDARY OUTCOMES:
Reduction of thyroid hormone overtreatment, measured as proportion of patients who had their TSH normalized. | 6 months post-enrollment
  Reduction in thyroid hormone overtreatment will be measured via EMR based on serum TSH in the normal range (=>0.5-6 mIU/L). We will assess TSH as a continuous variable and as a categorical variable (<0.5, 0.5-6, >6 mIU/L) to also delineate unintended TSH above the upper limit of normal.
Provider-reported knowledge | 6 months post-enrollment
  Assessed via surveys by provider report and defined as the composite score obtained from 4 items with response categories ranging from low to high (5-point Likert scale; 1: low to 5: high); higher scores indicate increased knowledge.
Provider-reported intent to deprescribe | 6 months post-enrollment
  Assessed via surveys by provider report (single item) with response categories ranging from low to high (5-point Likert scale; 1: very unlikely to 5: very likely).
Provider-reported self-efficacy | 6 months post-enrollment
  Assessed via provider surveys using the 9-item validated deprescribing self-efficacy survey designed to gain a better understanding of how providers rate their self-efficacy in deprescribing medications in their older adult patients (scale 0-100; higher scores indicate higher self-efficacy).
Patient-reported discussion of deprescribing with provider | 3-6 months post-enrollment
  Assessed via patient surveys by patient report and analyzed as a binary variable (yes/no).
Patient-reported knowledge | 3-6 months post-enrollment
  Assessed by patient surveys and will be defined as the percentage of correct answers (range 0-100%) from four questions regarding thyroid hormone therapy in older adults (true/false), where higher percentages indicate increased knowledge.
Patient-reported attitudes towards deprescribing | 3-6 months post-enrollment
  Assessed via patient surveys using the validated 22-item Revised Patients' Attitudes Towards Deprescribing (rPATD) questionnaire [subscales: perceived burden of medication taking, concerns about stopping the medication, belief in appropriateness of medication use (harms / benefits), level of involvement / knowledge of medications] and global questions. Questions pertaining to the burden, concerns about stopping, involvement in treatment, and global questions are scored such that a higher total score indicates a greater burden, concern, involvement, or agreement with global questions (5= strongly agree, 4= agree, 3= unsure, 2=disagree, 1= strongly disagree). Questions regarding the appropriateness factor were scored in reverse. In that case, a higher score indicates participants' belief in the appropriateness of their medications.
Patient-reported beliefs about medicines | 3-6 months post-enrollment
  Assessed via patient surveys using the validated 18-item Beliefs about Medicines Questionnaire (BMQ), with each item scored on a 5-point Likert scale (5= strongly agree, 4= agree, 3= unsure, 2=disagree, 1= strongly disagree). The BMQ is divided into BMQ-General (sub-scales: overuse and harm) and BMQ-Specific (subscales: necessity and concerns). Higher scores in the BMQ-General subscales indicate an overall negative perception of medications. Higher scores in the BMQ-Specific necessity subscale are indicative of a patient's need to adhere to medication to maintain health, while higher scores in the BMQ-Specific concerns subscale represent the notion that adverse reactions are potentially harmful when taking medication on a regular basis.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Papaleontiou, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
The researchers will make the de-identified data available to researchers upon reasonable request via email to the study PI at the conclusion of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For 5 years following publication
Access Criteria: Researchers